CLINICAL TRIAL: NCT05872477
Title: Promoting Repigmentation After Epidermal Cell Suspension Grafting and preVENTing the Loss of Melanocytes Using Topical Ruxolitinib for Vitiligo in Resistant Areas. Prospective Monocentric Interventional Study With Blinded Evaluation
Brief Title: Promoting Repigmentation After Epidermal Cell Suspension Grafting and preVENTing the Loss of Melanocytes Using Topical Ruxolitinib for Vitiligo in Resistant Areas
Acronym: PREVENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-PP-16
Record Dates: First submitted 2023-04-17; First posted 2023-05-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: There will be 2 arms with intra individual comparison. Each grafted side of the body will be randomly assigned to receive twice daily application of topical 1.5% ruxolitinib cream (Group A) or twice daily application of placebo cream (Group B). After 3 months, both sides will be treated by twice daily applications of topical ruxolitinib for 3 additional months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group treatment (Experimental): There will be 2 arms with intra individual comparison. After 7 days the dressing will be removed. Each grafted side of the body will be randomly assigned to receive twice daily application of topical 1.5% ruxolitinib cream After 3 months, both sides will be treated by twice daily applications of topical ruxolitinib for 3 additional months.
  Interventions: Drug: Ruxolitinib Topical
- group placebo (Placebo Comparator): Each grafted side of the body will be randomly assigned to receive twice daily application of placebo cream (Group B).
  After 3 months, both sides will be treated by twice daily applications of topical ruxolitinib for 3 additional months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib Topical — There will be 2 arms with intra individual comparison. Both groups will receive epidermal cell suspension (provided by Cutiss®). After 7 days the dressing will be removed. Each grafted side of the body will be randomly assigned to receive twice daily application of topical 1.5% ruxolitinib cream (Group A) or twice daily application of placebo cream (Group B). After 3 months, both sides will be treated by twice daily applications of topical ruxolitinib for 3 additional months.
  Arms: Group treatment
Drug: Placebo — There will be 2 arms with intra individual comparison. Both groups will receive epidermal cell suspension (provided by Cutiss®). After 7 days the dressing will be removed. Each grafted side of the body will be randomly assigned to receive twice daily application of topical 1.5% ruxolitinib cream (Group A) or twice daily application of placebo cream (Group B). After 3 months, both sides will be treated by twice daily applications of topical ruxolitinib for 3 additional months.
  Arms: group placebo

SUMMARY:
Medical approaches remain the gold standard treatment for non-segmental forms of vitiligo. Topical ruxolitinib cream has demonstrated its efficacy and good tolerance for treating vitiligo. While about 30% of patients will achieve at least 90% of repigmentation on the face after 1 year of treatment, some locations on the body, such as hands, feet, bony prominences remain highly challenging, and most patients won't get satisfactory repigmentation on those areas despite months of application of topical treatments, even when combined with UV. The poor rate of repigmentation in these locations are probably explained by the difficulty to stimulate the differentiation and proliferation of melanocytes stem cells in those areas. To study the efficacy at 3 months of epidermal cell suspension grafting followed by twice daily applications topical 1.5% ruxolitinib cream compared to epidermal cell suspension grafting followed by placebo in vitiligo resistant areas.There will be 2 arms with intra individual comparison. Both groups will receive epidermal cell suspension (provided by Cutiss®). After 7 days the dressing will be removed. Each grafted side of the body will be randomly assigned to receive twice daily application of topical 1.5% ruxolitinib cream (Group A) or twice daily application of placebo cream (Group B). After 3 months, both sides will be treated by twice daily applications of topical ruxolitinib for 3 additional months.There will be 8 visits in total during the 7 months duration for each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with non-segmental vitiligo.
2. ≥ 18 and <80 years.
3. At least one pair bilateral of stable vitiligo lesions with a surface >2cm² and < 20cm², located outside the face unresponsive to medical treatment
4. For women of child-bearing age, an effective contraception (estroprogestative pill, contraceptive implant, IUD, condoms or tubal ligation) should be used for more than one month before the inclusion in the study. A urine pregnancy test (βHCG in urines) will be performed.
5. Affiliation to a social security system
6. Signed informed consent
7. Participants who agree to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit.

Exclusion Criteria:

1. Pregnant or breast-feeding women. Or women who plan to get pregnant during the study duration.
2. Segmental or mixed vitiligo
3. Vitiligo lesions located only on face, feet, or fingers. (dorsum of the hand accepted).
4. Concomitant use of topical or systemic immunosuppressive medication or steroids
5. Previous treatment with topical ruxolitinib cream or any systemic JAK inhibitor
6. Areas that have already received surgical grafting
7. Patients suffering from photodermatosis or taking photosensitive drugs
8. Medical history of hypertrophic scars or keloids
9. Medical history of skin cancer on the site to be treated
10. Allergy to ruxolitinib cream, xylocaine or hyaluronic acid or trypsin (Viticell® must not be utilised with patients who are hypersensitive to hyaluronic acid or trypsin)
11. Active infection
12. Patients with thromboembolic risk
13. Any dermatosis located on the treated site that could interfere with the evaluation of the treatment
14. Vulnerable people: pregnant or breast-feeding women, minors, adult under guardianship or deprived of freedom
15. Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation
16. Participants with active acute bacterial, fungal, or viral skin infection within 1 week before baseline;
17. Participants with concurrent malignant disease or a history of that in the 5 years preceding the baseline visit except for adequately treated non metastatic malignancies;
18. Participants with current and/or history of liver disease, including known hepatitis B or C, with hepatic or biliary abnormalities;
19. Participants with current and/or history of tuberculosis;
20. Participants who have used depigmentation treatments for past treatment of vitiligo or other pigmented areas.
21. Patient under guardianship or curatorship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Repigmentation of the target area | At three months and visit inclusion.
  The primary objective will be assessed using the depigmentation of the target lesion. A drawing of the target lesions will be done at V1 (week 0), V5 (week 12) and V6 (wk24). Repigmentation of the target area will be calculated using Image J software in order to have an objective measurement of the response. We will define success as a repigmentation ≥50%, repigmentation being define as the difference of depigmentation between M3 and M0.

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided